CLINICAL TRIAL: NCT02422693
Title: Aquatic Exercises Versus Aquatic Exercises Associated to Deep Water-running for Patients With Chronic Low Back Pain: Randomized Controlled Trial
Brief Title: Aquatic Exercises for Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Collaborators: Ministry of Health, Brazil (Other Government); Fundação Araucária (Other)
Responsible Party: Principal Investigator, Jefferson Rosa Cardoso, PT, PhD, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: # 04/2012
Record Dates: First submitted 2015-04-06; First posted 2015-04-21 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Chronic Low Back Pain
Keywords: hydrotherapy; aquatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquatic exercises (Experimental): Warm-up, lumbar mobilization, stretching and relaxation. 3x-week (9 weeks), indoor pool, 32o.C/89.6o.F.
  Interventions: Other: Aquatic Exercises
- Aquatic exercises + Deep-water running (Active Comparator): Same as AEG with addition of 20 minutes of running without touch the ground, 3x-week (9 weeks), indoor pool, 30o.C/86o.F.
  Interventions: Other: Aquatic Exercises; Other: Deep-water running

INTERVENTIONS:
Other: Aquatic Exercises — Exercises performed in the water.
  Other Names: Aquatic Physical Therapy
Other: Deep-water running — It is a non-impact form of running executed in place in (higher than 2 meters) the water wearing a flotation belt. Heart rate is controlled by heart rate watch
  Arms: Aquatic exercises + Deep-water running

SUMMARY:
The goal of this study is to compare the effect of aquatic exercises (AEG) to the aquatic exercises plus aerobic training (deep-water running) (AEDWRG) on functional status and pain in patients with specific chronic low back pain.

DETAILED DESCRIPTION:
In general, the population will have at least one episode of low back pain during their lifetime, with recurrence in most cases. Several treatments have been proposed for these patients and the evidence is still not clear about the effectiveness of aquatic exercises when compared to other modalities of exercises in the water. This study will be a randomized controlled trial following the Consort-Statement principles. The subjects, aged between 20 and 50 years, after signing the informed consent will be randomly allocated to one group treatment: aquatic exercises (AEG) or aquatic exercises associated to deep-water running (AEDWRG). The duration of the protocol will be set at 12 weeks, 3x-week.

ELIGIBILITY:
Inclusion Criteria:

* Exclusive diagnosis of chronic low back pain (more than 12 weeks)

Exclusion Criteria:

* Central nervous system disease
* Pregnant
* Fear of water

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2017-01-29 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
Change in Roland-Morris Questionnaire | baseline and 9 weeks
  Functionality

SECONDARY OUTCOMES:
Change in Pain status | baseline and 9 weeks
  Pain

CONTACTS AND LOCATIONS:
Overall Officials: Jefferson R Cardoso, PT, PhD, Principal Investigator — Universidade Estadual de Londrina
Locations (1):
- Aquatic Physical Therapy Center "Paulo A. Seibert", Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No